CLINICAL TRIAL: NCT07113028
Title: Comparison of the Effectiveness of Conventional and Pulse Radiofrequency Therapy in Advanced Knee Osteoarthritis in Elderly Patients: An Observational Study
Acronym: pain
Status: Active, not recruiting | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Altun, pain specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Radiofrequency, knee pain
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Radiofrequency Ablation; Knee Arthritis Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Comparison of the Effectiveness of Conventional and Pulsed Radiofrequency Treatment in Advanced Knee

SUMMARY:
Knee osteoarthritis (OA) is a very common joint disease, causing pain and loss of function. Osteoarthritis, including knee OA, is a significant cause of morbidity and disability in older adults and negatively impacts the functionality of individuals over the age of 65. When non-invasive treatments such as medical therapy, physical therapy, and rehabilitation fail to provide adequate pain control, intra-articular injections, geniculate nerve blocks, radiofrequency ablation, and surgical treatments are considered.

Genicular nerve blocks provide short-term pain relief in knee osteoarthritis . Despite various conservative treatments, many patients with chronic knee OA experience severe knee pain before total knee arthroplasty. Genicular nerve block (GNB) and radiofrequency ablation of the geniculate nerves have been shown to be effective in relieving pain and improving knee functionality in patients with chronic knee OA. Intra-articular corticosteroids are used in the treatment of knee OA to rapidly relieve pain, reduce pain within the first three months, and rapidly restore joint function . Both conventional and pulsed radiofrequency treatments have been effective in relieving pain and improving disability in patients with knee OA who have not responded to conservative treatment and have contraindications for surgery. Conventional radiofrequency therapy uses high-frequency alternating current to create thermal lesions. The thermal energy creates a zone of coagulative necrosis that includes the nerves that transmit and/or modulate pain sensation . In pulsed radiofrequency therapy, thermal tissue damage can be minimized by using pulsed high-voltage radiofrequency currents. This allows time for the heat to dissipate and generally maintains the tissue temperature near the electrode below the neurodestructive range. The mechanism by which pulsed radiofrequency provides clinical benefit is not fully understood. It appears to modulate signaling cascades, particularly in C fibers, without affecting nerve conduction in myelinated fibers . As an alternative to the thermal effects of conventional radiofrequency therapy, pulsed radiofrequency therapy has been noted to have fewer potential side effects .

In conclusion, the therapeutic effects of radiofrequency applications on improving pain and functional impairments due to knee osteoarthritis (KOA) have been demonstrated; however, the number of studies evaluating only elderly patients (aged 65 and over) is limited. Studies comparing conventional and pulsed radiofrequency treatments of the genicular nerves and evaluating their effects on geriatric parameters are limited. The primary objective of our study was to compare the effects of conventional and pulsed radiofrequency treatments of the genicular nerves under ultrasound guidance on knee pain and functional assessments in elderly patients, and the secondary objective was to determine their effects on geriatric assessments.

DETAILED DESCRIPTION:
The study will be conducted at the Department of Algology at Kanuni Sultan Süleyman Training and Research Hospital by retrospectively reviewing the medical records of patients aged 65 and over diagnosed with knee osteoarthritis who underwent conventional or pulsed radiofrequency (USG)-guided radiofrequency (RF) treatment of the genicular nerves between January 2023 and March 2024. The interventional procedure is performed under sterile conditions, with the patient monitored, supported below the knee, and in slight flexion, adhering to asepsis and antisepsis guidelines. The genicular nerves are visualized using ultrasound guidance, and radiofrequency treatment is administered in conventional or pulsed mode, followed by appropriate sensory and motor stimuli. Demographic data, height, weight, duration of symptoms, comorbidities, analgesic use, pre-treatment and post-treatment 1st and 3rd month Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Numeric Rating Scale-11 (NRS-11), Tinneti Balance, Tinneti gait and performance-oriented mobility assessment (POMA), and timed up and go test will be recorded from the patient files.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone ultrasound-guided genicular nerve RFT.
* Patients over the age of 65 who have a diagnosis of knee OA and who cannot achieve adequate pain palliation with conservative treatments.
* Patients with complete data to be scanned in their files.

Exclusion Criteria:-Patients who have received radiofrequency treatments other than those diagnosed with osteoarthritis

* Patients who have received intra-articular knee injections, PRP, or hyaluronic acid injections in the last 6 months
* Patients who have undergone knee replacement surgery
* Patients diagnosed with malignancy
* Patients who have received steroids for any reason in the last 6 months
* Patients with radicular pain
* Connective tissue diseases
* Serious neurological or psychiatric disorders
* Mental impairment that prevents adequate communication or cooperation Use of anticoagulant medications

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study will include 60 patients aged 45 years and over, diagnosed with Kellgren-Lawrence (KL) stage 3-4 knee osteoarthritis, who underwent ultrasound-guided geniculate radiofrequency (RFT) between January 2022 and January 2023 at the Algology Department of Kanuni Sultan Süleyman Training and Research Hospital. The minimum number of patients required to achieve a 10% difference (normal width = 4.5 + 0.4 mm), i.e., a difference of approximately 0.5 mm, was determined to be 30 (80% power, p<0.05). Considering the losses, the planned inclusion of 60 patients is planned.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale-11 (NRS-11): This is an 11-point scale used to describe pain. It is based solely on the patient's ability to perform activities of daily living and can be used for adults and children ages 10 and older. | 1 month

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities. Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC consists of five items for pain (score range 0-20), two items for stiffness (score range 0-8), and 17 items for functional limi | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Küçükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided